CLINICAL TRIAL: NCT00731588
Title: Red Blood Cell Survival Following Transfusion in Infants
Brief Title: Red Blood Cell (RBC) Survival Following Transfusion in Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John A Widness (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Thrasher Research Fund (Other)
Responsible Party: Sponsor-Investigator, John A Widness, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200710747; 2P01HL046925 (NIH)
Record Dates: First submitted 2008-08-05; First posted 2008-08-11 (Estimated); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Neonatal Anemia
MeSH Terms: conditions — Anemia, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PPG1A - Adults (Experimental): Phase I completed: Healthy male and post-menopausal female volunteers between the ages of 18 and 65. Volunteers must not have donated blood in the previous 8 weeks.
  Interventions: Biological: Transfused Biotin RBCs - Adults Phase I
- PPG1B - Infants (Experimental): Phase II in progress: Newborns >= 24 weeks gestation who are patients in the Neonatal Intensive Care Unit at the University of Iowa Hospitals and Clinics that are being treated with the expectation of survival.
  Interventions: Biological: Transfused Biotin RBCs - Infants Phase II; Biological: Transfused Biotin RBCs - Infants Phase III

INTERVENTIONS:
Biological: Transfused Biotin RBCs - Adults Phase I — A 3 mL venous blood sample is obtained. 250 mL of blood will be drawn to a blood collection bag containing the anticoagulant CPD. Separate equal volumes of RBCs are labeled with up to five different densities of biotin. The biotinylated RBCs are resuspended in autologous plasma to achieve a 60 to 70% hematocrit. An IV is inserted for the reinfusion of the biotinylated RBCs. Three mL aliquots of blood are sampled at 5, 10, 20, and 60 minutes after infusion. The subject returns ~24 hours and 3 days after the RBC infusion to obtain a 3 mL venous blood sample. Subjects return for weekly 3 mL blood sampling.
  Arms: PPG1A - Adults
Biological: Transfused Biotin RBCs - Infants Phase II — After the infant's clinical care team decides that a RBC transfusion is needed, a 15mL/kilogram of body weight is ordered. Transfusion will be given in 2 parts: 1) approximately 80% of the total transfusion to be transfused over 3-4 hours and 2) approximately 20% of the total transfusion will be marked with biotin to be transfused upon completion of the first part. The bedside nurse maintains constant observation of the infant as appropriate for the infant's condition, assessing for signs and symptoms of a transfusion reaction.
  Arms: PPG1B - Infants
Biological: Transfused Biotin RBCs - Infants Phase III — Phase III (infants) to be determined upon completion of Phase II (infants).
  Arms: PPG1B - Infants

SUMMARY:
OUR OVERALL HYPOTHESIS is that post-transfusion survival of allogeneic and autologous RBCs can be accurately quantified in anemic human infants using biotin-labeled RBCs combined with mathematical modeling that adjusts for confounding factors commonly encountered in neonates. These confounding factors include 1) dilution of labeled RBC as a result of growth stimulated erythropoiesis, anemia stimulated erythropoiesis, and blood transfusion; 2) loss of labeled RBC due to laboratory phlebotomy; and 3) variable RBC life spans resulting from RBCs having been produced at different developmental periods and under varying rates of erythropoiesis. In contrast to infants, adjustment for these factors is not necessary in healthy adults under conditions of steady state erythropoiesis. Instead in adults, RBC survival is typified by a linear decline in concentration of labeled RBCs over time. When this line is extrapolated to zero concentration, the intercept with the time axis represents the mean potential lifespan (MPL) of RBCs. (<7 d) and stored (>21 d) allogeneic adult RBCs transfused in the same infant.

DETAILED DESCRIPTION:
Phase I: Includes only Aim #1 from Thrasher Foundation Grant in which adult subjects will be studied.

SPECIFIC AIM #1 (Thrasher Foundation Grant): To develop in vitro and validate in vivo in adult humans and anemic infants the capability of biotinylating RBCs at up to 5 discrete densities for simultaneously determining RBC kinetics of multiple, distinct RBC populations. This requires expansion of the RBC biotin labeling technology we have previously developed. After refinement, the method will be applied in the subsequent aims conducted in anemic infants receiving clinically ordered RBC transfusions.

As suggested by our previous RBC survival studies, we anticipate that the heaviest biotin labeling will alter the intrinsic RBC structural properties of RBCs, shortening their long term survival. The in vitro and in vivo validation studies we propose in adults are necessary because the conditions for reproducibly obtaining discrete RBC biotin densities at appropriate, closely spaced intervals have not been conclusively worked out, nor have we determined empirically which of the five densities will not artifactually shorten long-term RBC survival. We can use the lighter densities for RBC survival measurements and the heavier densities for the simultaneous RBC volume measurements needed to account for RBC volume increases caused by growth. It is important to perform these feasibility studies in both adults and infants because of the vastly different physiologic states, ie, normal, healthy adults are in steady state erythropoiesis while critically ill, anemic infants experience multiple clinical circumstances which perturb RBC survival, eg, growth, phlebotomy, intervening transfusion, etc.

In addition to the biotin labeling of RBC method, the "differential agglutination, antigenic method" using flow cytometry will be applied for infants receiving allogeneic RBC transfusions. The results of the two methods will be compared with one another. The differential agglutination method utilizes differences in the RBC surface antigens between the donor and the recipient for determining short- and long-term RBC survival. Genotyping results of adult donor and the infant recipient RBC antigens (performed at the Mississippi Valley Regional Blood Center) permits identification of minor blood group differences between donor and recipient RBCs so that appropriately labeled minor RBC antibodies (available commercially and used by blood banks for minor blood group RBC typing) can be used in flow cytometric determination of RBC survival. RBC survival determined for each of the biotin labels and for the RBC antigenic differences will all be compared among one other. The differential agglutination/antigen method will considered the "gold standard" as the RBCs are labeled ex-vivo, AFTER the RBC transfusion, thus without modifying the RBC membrane surface proteins as biotinylation does. Our hypothesis is that the addition of too much biotin can lead to artifactually shortened in vivo RBC survival, but that lower doses of biotin to not. By also including the differential agglutination/antigen method RBC survival results, we will be able to better validate our multi-density biotin hypothesis.

Our overall objective in this research is to improve red blood cell (RBC) transfusion practices for anemic, critically ill infants. This project has received support from two granting agencies: 1) The Thrasher Foundation, entitled, "Red Blood Cell Recovery and Survival Following Transfusion in Infants;" and 2) NIH PPG Grant P01 HL046925, Project 1 entitled, "Red Blood Cell Survival Following Transfusion In Infants." Abstracts for both are included below. This project will be completed in two phases:

Phase I includes studies of autologous biotinylated RBCs transfused into normal, health adult human volunteers (see Specific Aim #1 in Thrasher Foundation Abstract below); and

Phase II includes studies of infants requiring physician order red blood cell transfusions (see Specific Aims #2, #3, and #4 in Thrasher Foundation Abstract below; and see Specific Aim #4 in NIH which is included in its entirety in the three Thrasher Grant specific aims).

The Phase I studies are completed and we are no longer enrolling adults. We are enrolling infants for Phase II studies. We are adding these phases sequentially based on the recommendation of Martha Jones at the time our proposal was first submitted to the IRB. We have applied the knowledge we have gained from the Phase I studies in adult subject volunteers to make modifications of our study design for Phase II to be performed in infant study subjects receiving clinically ordered RBC transfusions. At the end of Phase II, justification for including a new, comparison "gold standard" method for determining RBC survival in infants (the "differential agglutination, antigenic method") is included. We have completed enrollment of all adult subjects for phase I.

ABSTRACT I (FOR THRASHER FOUNDATION GRANT)

Background:

Anemic, critically ill newborn infants are among the most frequently transfused groups of patients in the US. An estimated 130,000 infants annually receive approximately 1,000,000 RBC transfusions. Unlike adults, important data are lacking regarding the transfusion product for optimal RBC survival in infants. Contributing to this lack are two major recent changes in neonatal blood banking and transfusion practices. These are 1) the use of transfused adult donor blood stored for up to the 42 day FDA limit instead of only using blood stored for less than 7 days as had been done previously; and 2) potential use of the infant's own blood harvested from the placenta to avoid the risks of viral infections and immune transfusion reactions from donor blood. Unfortunately, there are no definitive infant studies that address these changes by directly measuring RBC survival. Such infant studies have been hampered by technical problems. Specifically, RBC survival data must be adjusted for growth, laboratory phlebotomy loss, and intervening additional RBC transfusions but in practice have not. Moreover, safety issues have precluded many infant RBC survival studies (eg, exposure to 51Cr radioactivity and removal of too much blood from today's tiny, premature infants). Indeed, prior to 1970 (the end of using 51Cr as a RBC label in infant RBC survival studies), infants weighing less than 1,500 g at birth did not often survive, and RBC survival data do not exist for today's smallest, most frequently transfused infants whose birth weights are 500-1,000 g.

Specific Aims:

Specific Aim #1: To develop in vitro and validate in vivo in adults the capability for biotinylating RBCs at up to 5 discrete densities that are measurable by flow cytometry. These five RBC biotin density labels will be used in Specific Aims #2, 3, and 4 to simultaneously determine RBC survival of multiple, distinct populations of transfused RBCs in premature infants.

Specific Aim #2. To determine whether RBC survival of donor and placental RBCs are significantly longer when adjusted by mathematical modeling. We anticipate that the unmodeled values substantially underestimate RBC survival.

Specific Aim #3. To compare long-term RBC survival results for transfused adult donor and fetal/placental RBCs in anemic newborn infants. We anticipate that more rapid growth in fetuses will result in greater stress erythropoiesis leading to intrinsic RBC "defects" and shortened RBC survival compared to adult donor RBCs.

Specific Aim #4. To quantify the effects of storage on model adjusted RBC survival of adult donor RBCs transfused into newborn infants. We anticipate that storage of donor RBCs will not alter RBC survival.

Study Design:

The studies proposed here build on biotinylation and mathematical modeling methods that our research group has developed for accurately measuring RBC survival without exposing the infant to radioactivity. The biotin RBC labeling method is well suited to newborn infants because it permits the simultaneous tracking of multiple RBC populations on <10 µL blood. Survival of RBCs labeled at multiple biotin densities will be quantified using the standard RBC survival parameters, ie, post-transfusion short-term 24 h RBC recovery and long-term modeled RBC survival, ie, until 50 and 100% of biotin-labeled RBCs have disappeared from the circulation. The latter two measurements will be calculated using the required mathematical adjustments for growth, laboratory phlebotomy loss, and intervening RBC transfusions.

Only Specific Aim #4 in the Thrasher Foundation Abstract involves human infant study subjects. Specific Aim #4) USE THE RBC BIOTINYLATION AND MATHEMATICAL MODELING METHODOLOGIES VALIDATED IN ADULT SHEEP AND NEWBORN LAMBS TO ACCURATELY MEASURE POST-TRANSFUSION RBC KINETICS IN ANEMIC NEWBORN INFANTS TRANSFUSED WITH FRESH AUTOLOGOUS, FRESH ALLOGENEIC AND STORED ALLOGENEIC RBCS. The use of biotin, a non-toxic, non-radioactive B vitamin, to distinguish among different RBC populations simultaneously by flow cytometry is critical for accomplishing our aims and holds clear advantages over other RBC labeling methods in both safety and accuracy. In utilizing the four Specific Aims to achieve our goal of establishing more effective transfusion practices by identifying the optimal RBC transfusion product for use in anemic INFANTS.

ELIGIBILITY:
Adult Study:

Inclusion Criteria:

* Males or post-menopausal females
* 18-65 years of age.
* Weight >110 lbs.
* Healthy- the subject feels well and can perform normal activities.
* Hemoglobin at or above 12.5 g/dL or hematocrit at or above 38%.

  * Note: Members of the research team that are not supervised or under the employee of the PI may participate in the study.

Exclusion Criteria:

* Presence of chronic illness unless the subject is being treated and the condition is under control.
* Consumption of biotin supplements or raw eggs.
* Premenopausal women.
* Blood donation in the previous 8 weeks (single donation) or 16 weeks (double red cell donation).
* Blood loss in the previous 8 weeks due to epistaxis, gastrointestinal blood loss, trauma, significant diagnostic phlebotomy loss (i.e., > 30 mL total), or other significant bleeding
* Treatment with antibiotics within the last 7 days. Antibiotics for prevention of an infection or treatment of acne are not exclusion criteria.

  * Note: If study subjects experience any of these conditions associated with blood loss or donate any blood products, they will not be included in the primary analysis but will be replaced.

Infant Study:

MOTHERS FOR PLACENTAL BLOOD COLLECTION AND MOTHERS OF INFANT STUDY SUBJECTS

Inclusion Criteria:

1. >/= 24 weeks gestation
2. mothers who deliver through the birth canal or by c-section can be included in the study.

Exclusion Criteria:

1. Pregnant with fetus with major congenital anomaly.
2. Clinically suspected or documented maternal chorioamnionitis (This only applies to infant study subjects receiving autologous RBCs from the placenta).
3. Viral or bacterial infection (e.g. HIV, Hepatitis B, Hepatitis C, Primary Herpes, Tuberculosis) based on clinically available prenatal or postnatal test results in the mother's medical record. (This only applies to infant study subjects receiving autologous RBCs from the placenta.)
4. minor mothers (<18 years old) are excluded from the study.

INFANT STUDY SUBJECTS

Inclusion Criteria:

Newborns >/=24 weeks gestation who are patients in the Neonatal Intensive Care Unit (NICU) at UIHC that:

1) Are being treated with the expectation of survival.

Exclusion Criteria:

1. Difference of more than 5% in the percentage of HbF cells (measured by flow cytometry in the Widness lab) between blood harvested from the placenta and that from discarded neonatal blood in the first day of life and before the first neonatal blood transfusion. This is done to exclude the rare possibility of transfusing newborns with blood that is contaminated with a significant proportion of their mother's blood if a maternal-to-placenta bleed occurs after umbilical cord clamping is done. (This only applies to infant study subjects receiving autologous RBCs from the placenta.)
2. Need of emergent blood transfusion as determined by the subject's medical care team.
3. Hematological diseases (except for anemia associated with phlebotomy loss and prematurity)
4. Alloimmune hemolytic anemia, diffuse intravascular coagulation, and thrombosis.
5. Major congenital anomaly.
6. Sepsis with positive blood or spinal fluid culture.
7. Receiving treatment with erythropoietin (r-HuEPO) or cardiorespiratory bypass support (ECMO).
8. Overt clinical bleeding.

Ages: 1 Hour to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Widness, MD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Iowa, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mock DM, Matthews NI, Strauss RG, Burmeister LF, Schmidt R, Widness JA. Red blood cell volume can be independently determined in vitro using sheep and human red blood cells labeled at different densities of biotin. Transfusion. 2009 Jun;49(6):1178-85. doi: 10.1111/j.1537-2995.2009.02095.x. Epub 2009 Feb 10. PMID 19220818
- [Result] Mock DM, Matthews NI, Zhu S, Burmeister LF, Zimmerman MB, Strauss RG, Schmidt RL, Nalbant D, Cress GA, Widness JA. Red blood cell (RBC) volume can be independently determined in vivo in humans using RBCs labeled at different densities of biotin. Transfusion. 2011 Jan;51(1):148-57. doi: 10.1111/j.1537-2995.2010.02770.x. PMID 20630041
- [Result] Mock DM, Matthews NI, Zhu S, Strauss RG, Schmidt RL, Nalbant D, Cress GA, Widness JA. Red blood cell (RBC) survival determined in humans using RBCs labeled at multiple biotin densities. Transfusion. 2011 May;51(5):1047-57. doi: 10.1111/j.1537-2995.2010.02926.x. Epub 2010 Nov 9. PMID 21062290
- [Result] Mock DM, Lankford GL, Matthews NI, Burmeister LF, Kahn D, Widness JA, Strauss RG. Accelerated removal of antibody-coated red blood cells from the circulation is accurately tracked by a biotin label. Transfusion. 2012 May;52(5):1097-105. doi: 10.1111/j.1537-2995.2011.03397.x. Epub 2011 Oct 24. PMID 22023312
- [Result] Mock DM, Widness JA, Strauss RG, Franco RS. Posttransfusion red blood cell (RBC) survival determined using biotin-labeled RBCs has distinct advantages over labeling with (51) Cr. Transfusion. 2012 Jul;52(7):1596-8. doi: 10.1111/j.1537-2995.2012.03588.x. No abstract available. PMID 22780899
- [Result] Nalbant D, Bhandary P, Matthews NI, Schmidt RL, Bogusiewicz A, Cress GA, Zimmerman MB, Strauss RG, Mock DM, Widness JA. Comparison of multiple red cell volume methods performed concurrently in premature infants following allogeneic transfusion. Pediatr Res. 2013 Nov;74(5):592-600. doi: 10.1038/pr.2013.143. Epub 2013 Sep 3. PMID 24088873
- [Result] Widness JA, Nalbant D, Matthews NI, Strauss RG, Schmidt RL, Cress GA, Zimmerman MB, Mock DM. Tracking donor RBC survival in premature infants: agreement of multiple populations of biotin-labeled RBCs with Kidd antigen-mismatched RBCs. Pediatr Res. 2013 Dec;74(6):689-97. doi: 10.1038/pr.2013.163. Epub 2013 Sep 4. PMID 24108188
- [Result] Widness JA, Kuruvilla DJ, Mock DM, Matthews NI, Nalbant D, Cress GA, Schmidt RL, Strauss RG, Zimmerman MB, Veng-Pedersen P. Autologous Infant and Allogeneic Adult Red Cells Demonstrate Similar Concurrent Post-Transfusion Survival in Very Low Birth Weight Neonates. J Pediatr. 2015 Nov;167(5):1001-6. doi: 10.1016/j.jpeds.2015.08.028. Epub 2015 Sep 9. PMID 26363547
- [Result] Schmidt RL, Mock DM, Franco RS, Cohen RM, North AK, Cancelas JA, Geisen C, Strauss RG, Vlaar AP, Nalbant D, Widness JA. Antibodies to biotinylated red blood cells in adults and infants: improved detection, partial characterization, and dependence on red blood cell-biotin dose. Transfusion. 2017 Jun;57(6):1488-1496. doi: 10.1111/trf.14075. Epub 2017 Mar 5. PMID 28261808
- [Derived] Nalbant D, Cancelas JA, Mock DM, Kyosseva SV, Schmidt RL, Cress GA, Zimmerman MB, Strauss RG, Widness JA. In premature infants there is no decrease in 24-hour posttransfusion allogeneic red blood cell recovery after 42 days of storage. Transfusion. 2018 Feb;58(2):352-358. doi: 10.1111/trf.14396. Epub 2017 Nov 29. PMID 29193118

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some infants (actually the mothers were asked for consent for their infants) were enrolled before birth and then after birth were found to be ineligible. No cord blood was available in some cases and thus could not be studied.
Period: Overall Study
Arm/Group | PPG1A - Adults | PPG1B - Infants
Started | 9 | 95
Completed | 9 | 53
Not Completed | 0 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PPG1A - Adults | PPG1B - Infants | Total
Number analyzed (Participants) | 9 | 53 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 53 | 53
  Between 18 and 65 years | 9 | 0 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 32 | 38
  Male | 3 | 21 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 9 | 47 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 53 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Discrete Biotinylated RBC Densities (up to 5 Discrete Densities) That Can be Accurately Measured by Flow Cytometry, i.e., Without Overlap.
Description: The biotin-labeled RBCs that were studied were: 2, 6, 18, 54, and 162 µg NHS-biotinylating reagent per mL of packed RBCs. Here we report the number of discrete biotin densities without overlap as determined in vitro.
Time Frame: from day of blood draw this can be accomplished in 4 hours
Population: These were representative samples studied in vitro from infants and adults
Measure: Number; unit: flow cytometry RBC discrete peaks
Arm/Group | PPG1A - Adults | PPG1B - Infants
Number analyzed (Participants) | 3 | 3
flow cytometry RBC discrete peaks | 5 | 5

2. Primary Outcome: RBC Survival (Life Span) in Days of Multiple, Distinct BioRBC Density Populations of Transfused Autologous RBCs in Adults and Premature Infants.
Description: Using flow cytometry was measured for each RBC biotin density in days as determined when RBC measurement was no longer detectable.
Time Frame: for up to 5 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PPG1A - Adults | PPG1B - Infants
Number analyzed (Participants) | 9 | 53
days
  BioRBC 2 µg/mL | NA (NA) — Adults were never studied at the 2 µg/mL BioRBC density. The is because our protocol did not allow for normal adults to be studied at this BioRBC density. | 60 (20)
  BioRBC 6 µg/mL | 120 (10) | 60 (20)
  BioRBC 18 µg/mL | 120 (10) | 60 (20)
  BioRBC 54 µg/mL | 95 (10) | 60 (20)
  BioRBC 162 µg/mL | 80 (10) | NA (NA) — This was not tested infants because of prior results in adults.

3. Primary Outcome: RBC Survival (Life Span) in Days of Multiple, Distinct BioRBC Density Populations of Transfused Allogeneic RBCs in Premature Infants.
Description: as for outcome 2
Time Frame: for up to 4 months
Population: This only applies to infants since no adults received allogeneic biotin labeled RBC
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PPG1B - Infants
Number analyzed (Participants) | 40
days
  BioRBC 2 µg/mL | 60 (20)
  BioRBC 6 µg/mL | 60 (20)
  BioRBC 18 µg/mL | 60 (20)
  BioRBC 54 µg/mL | 60 (20)

4. Secondary Outcome: Number of Participants With Positive Antibody Screen in Response to Biotin-labeled RBCs.
Description: IgG gel card agglutination test that was developed in our laboratory
Time Frame: 4 to 5 mo post transfusion of biotin RBCs
Measure: Count of Participants; unit: Participants
Arm/Group | PPG1A - Adults | PPG1B - Infants
Number analyzed (Participants) | 9 | 53
Participants | 3 | 0

5. Secondary Outcome: Survival of Allogeneic RBCs in Days as Measured by the Antigenic Method Using Flow Cytometry for Comparison With BioRBC in Premature Infants
Time Frame: 4 months
Population: Only applies to allogeneic RBCs and all infants did not have autologous transfusions
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PPG1B - Infants
Number analyzed (Participants) | 40
days | 70 (20)

ADVERSE EVENTS:
Time Frame: 5 months for adults, 4 months for infants
Arm/Group | PPG1A - Adults | PPG1B - Infants
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/53
Other Adverse Events (participants affected / at risk) | 0/9 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT00731588/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT00731588/SAP_001.pdf